CLINICAL TRIAL: NCT01042613
Title: A Comparison of the Success Rate Of Cannulation Between The Accuvein Apparatus And Standard Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACVEIN
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-11

CONDITIONS: Cannulation
Keywords: AccuVein AV300 device;; Intravenous cannulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Research participants are randomly assigned into group A (Accuvein AV300 assisted intravenous catheter insertion)
  Interventions: Procedure: Cannulation using Accuvein device
- Group B (Other): (standard technique of insertion of the intravenous cannula)
  Interventions: Procedure: Standard Cannulation method

INTERVENTIONS:
Procedure: Cannulation using Accuvein device — If the research participant has been randomized to the AV300 device group A, then intravenous cannulation will be attempted using the AV300 device following manufacturer's instructions by four anesthesiologists.
  Arms: Group A
Procedure: Standard Cannulation method — If the research participant has been randomized to the standard treatment group B then cannulation will be attempted in the standard manner. A research team member will time cannulation access for all participants. Participation ends once successful cannulation is achieved or when a maximum of 4 skin punctures have been made.
  Arms: Group B

SUMMARY:
1. This study will compare the first attempt success rate of cannulation in research participants randomized to using a new FDA approved AccuVein AV300 device for intravenous access with research participants randomized to standard cannulation methods.
2. This study will assess if insertion of intravenous cannula is faster when intravenous access is assisted by the AccuVein AV300 device as compared to the standard technique.
3. This study will assess if the number of skin punctures is fewer when intravenous access is assisted by the AccuVein AV300 device as compared to the standard technique.

DETAILED DESCRIPTION:
Patients agreeing to participate in this study will be randomized to one of two groups for intravenous access. One group will use the standard cannulation method and the other group will use the new FDA approved AccuVein AV300 device for cannulation.

After pre-anesthetic evaluation, the research participant will be brought to the operating room or magnetic resonance imaging (MRI) Suite and standard monitoring will be applied (EKG, SpO2, BP) if tolerated. Anesthesia will be induced via a face mask with sevoflurane in 100% O2. When the supervising anesthesiologist deems it appropriate, attempt at cannulation will begin.

A tourniquet will be applied. A 22-gauge cannula will be used. Randomization will take place before the patient is taken back to the Operating Room or MRI Suite. If the research participant has been randomized to the standard treatment group then cannulation will be attempted in the standard manner. If the research participant has been randomized to the AV300 device group then intravenous cannulation will be attempted using the AV300 device following the manufacturer's instructions.

A research team member will time cannulation access for all participants. Participation ends once successful cannulation is achieved or when a maximum of 4 skin punctures have been made.

Only the study coordinator will know which randomization group the patient has been assigned. Once the anesthesiologist has determined a potential IV access site, s/he will be informed to which group the patient was assigned. If the parent/guardian requests, s/he will be told after the procedure to which group the child was randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children under 18 years of age.
2. American Society of Anesthesiologist (ASA) Physical Status I, II or III.
3. Patients undergoing elective surgery,examination under anesthesia,or MRI who do not have existing intravenous access.
4. Able to understand English.
5. Parent/guardian willing to sign consent.

Exclusion Criteria:

1. Existing intravenous access.
2. Malformations or infections at the potential site of insertion.
3. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
4. Need for emergency surgery.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Trujillo Huaccho, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 148 total patients were recruited at single institution (SJCRH) study between Jan 13, 2010, and March 03, 2011.
Pre-assignment Details: 148 total patients were enrolled on the study. The report is based on results for 146 patients. Two patients were excluded from this study. One patient was excluded due to MD's decision and the other patient was deemed to be inevaluable after study enrollment (cannula gauge other than 22 were used).
Groups:
- ACVein: Research participants are randomly assigned into group A (Accuvein AV300 assisted intravenous catheter insertion)
- Standard: (standard technique of insertion of the intravenous cannula)
Period: Overall Study
Arm/Group | ACVein | Standard
Started | 72 | 74
Completed | 72 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACVein | Standard | Total
Number analyzed (Participants) | 72 | 74 | 146
Age Continuous [Mean (Standard Deviation); unit: years] | 5.72 (3.72) | 5.37 (3.88) | 5.54 (3.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 43 | 78
  Male | 37 | 31 | 68

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate of Cannulation
Description: This study will compare the first attempt success rate of cannulation in research participants randomized to using a new FDA approved AccuVein AV300 device for intravenous access with research participants randomized to standard cannulation methods. There is one timepoint for outcome data collection and it is prior to cannulation. Success (yes) is defined as needle insertion into target vein.
Time Frame: At cannulation
Population: Patients (age 17 years or less) undergoing elective surgery or examination under anesthesia who do not have existing intravenous access.
Measure: Number; unit: Participants
Arm/Group | ACVein | Standard
Number analyzed (Participants) | 72 | 74
Participants
  Successful first attempt | 54 | 54
  Unsuccessful first attempt | 18 | 20
Statistical Analysis 1: Comparison: ACVein vs Standard; Test type: Superiority or Other; p = .851, Fisher Exact; Difference of the Binomial Proportions = .02

2. Secondary Outcome: Time Between Tourniquet Application and Successful Cannulation is Achieved or 4 Attempts Have Been Made (in Minutes).
Description: To assess if insertion of intravenous cannula is faster when intravenous access is assisted by the AccuVein AV 300 device as compared to the standard technique
Time Frame: At cannulation
Population: Of the 146 patients, two patients were excluded due to missing time records.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | ACVein | Standard
Number analyzed (Participants) | 71 | 73
Minutes | 1.48 (.97) | 1.26 (.84)
Statistical Analysis 1: Comparison: ACVein vs Standard; Test type: Superiority or Other; p = .105, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .22

3. Secondary Outcome: Number of Skin Punctures
Description: To assess if the number of skin punctures is fewer when intravenous access is assisted by the AccuVein AV300 device as compared to the standard technique
Time Frame: At cannulation
Measure: Mean (Standard Deviation); unit: Skin punctures
Arm/Group | ACVein | Standard
Number analyzed (Participants) | 72 | 74
Skin punctures | 1.33 (.75) | 1.26 (.62)
Statistical Analysis 1: Comparison: ACVein vs Standard; Test type: Superiority or Other; p = .8, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = .07

ADVERSE EVENTS:
Time Frame: 10 minutes per patient
Description: Enrollment was from January, 2010 through March, 2011. Patients were off study at completion of cannulation.
Arm/Group | ACVein | Standard
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/74
Other Adverse Events (participants affected / at risk) | 0/72 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes